CLINICAL TRIAL: NCT06233032
Title: Could Ephedrine Replace Dexmedetomidine for Prevention of Shivering in Women Undergoing Cesarean Section Under Spinal Anaesthesia
Brief Title: Could Ephedrine Replace Dexmedetomidine Fordexmedetomidine Prevention of Shivering in Women Undergoing Cesarean Section Under Spinal Anaesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Salah Kamal Salman, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Prevention of shivering
Record Dates: First submitted 2023-09-05; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-06

CONDITIONS: Prevention of Shivering With Spinal Anaesthesia
MeSH Terms: interventions — Ephedrine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E (Experimental)
  Interventions: Drug: Ephedrine
- Group D (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Ephedrine — Patient Will receive 6mg IV
  Arms: Group E
Drug: Dexmedetomidine — Patient Will receive 30mcg IV
  Arms: Group D

SUMMARY:
Could ephedrine replace dexamedetomidine for prevention of shivering in women undergoing Cesarean section Under spinal anaesthesia

DETAILED DESCRIPTION:
Shivering, rhythmic oscillatory movement of upper limbs, neck and jaw, is common during regional anesthesia with an incidence up to 56.7% of patients. Perioperative shivering is a commonly observed clinical problem well known to anesthesiologists caring for women undergoing a Cesarean delivery (CD). The median incidence of shivering in parturients having labour epidural analgesia or CD with epidural or spinal anesthesia has been estimated to be 52%.1 Severe shivering causes physiologic stress, interferes with patient monitors, and decreases the comfort and overall satisfaction of women during childbirth. Ephedrine well-known sympathomimetic agent, has been used to treat hypotension during regional anesthesia. It has antiemetic effect for short-term . Ephedrine maintained hemodynamics and minimized decrease of the core temperature when given by an intravenous infusion during spine surgery under general anesthesia . Dexmedetomidine, a selective a-2 agonist, was introduced in clinical practice in the United States in 1999. It is approved by Health Canada as a short-term sedative for mechanically ventilated adult patients in the intensive care unit and sedation of non-intubated patients prior to and/or during surgical procedures. It has since been approved and is widely used in pediatric populations and for procedural sedation of non-intubated patients.9 Nevertheless, the clinical use of dexmedetomidine has expanded to various off-label uses. In obstetrical anesthesia, it has been used as part of multi-modal intravenous labour and post-CD analgesia,10-13 as a neuraxial adjunct in the epidural space for labour,14 and intrathecally for shivering prevention during CD

ELIGIBILITY:
Inclusion Criteria:

* Adult female from 18 to 35 yrs
* uncomplicated pregnancy for elective cesarean delivery

Exclusion Criteria:

* patient refusal
* allergy to the drug
* contraindications of spinal anaesthesia
* patients with DM or thyroid disorders

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Prevention of shivering during spinal anaesthesia in cesarean delivery .Intensity of shivering assessed using five point scale | 45min
  one hundred Pts will be included in this study .
  1. fifty patients will receive Ephedrine 6 mg IV bolus before spinal block.
  2. fifty patients will be receive 30 microgram IV bolus before spinal block

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No